CLINICAL TRIAL: NCT05051007
Title: Comparison of the Hemodynamic Effects of Opioid-based Versus Lidocaine-based Induction of Anesthesia With Propofol in Elderly: A Randomized Controlled Study
Brief Title: Opioid-based Versus Lidocaine-based Induction of Anesthesia With Propofol in Elderly
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Maha Mostafa Ahmad, MD, Principal Investigator, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MD-239-2021
Record Dates: First submitted 2021-09-10; First posted 2021-09-21 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Postinduction Hypotension; Elderly
MeSH Terms: interventions — Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fentanyl group (Active Comparator)
  Interventions: Drug: fentanyl
- lidocaine group (Active Comparator)
  Interventions: Drug: Lidocaine IV

INTERVENTIONS:
Drug: fentanyl — patients will receive 1 mcg/kg of fentanyl (the drug will be diluted to 10 mcg/mL)
  Arms: fentanyl group
Drug: Lidocaine IV — patients will receive 1 mg/kg lidocaine (the drug will be diluted to10mg/mL)
  Arms: lidocaine group

SUMMARY:
Advances in the medical service and public health increased longevity; hence, more elderly patients (>65 years) are encountered by the anesthetists for variety of surgical interventions. Even with the absence of comorbidity, older patients represent a challenge to the anesthetist in comparison to the younger patients due to their limited physiologic reserve and their aberrant response to the varies perioperative medications.

Intraoperative hypotension increases the risk of postoperative kidney injury, myocardial injury, cerebral ischemia, and perioperative mortality. Postinduction hypotension is mainly caused by anesthetic drugs. Hence, developing a technique for induction of anesthesia that provide adequate hypnosis with stable hemodynamics during surgery is critical, especially for elderly patients. The elderly patients are at increased risk of post-induction hypotension due to increased drug sensitivity.

Propofol is the most commonly used drug for anesthesia induction; however, its use is usually associated with hypotension through vasodilation and direct myocardial depression. Opioid drugs are usually added as analgesics to propofol during induction of anesthesia. However, addition of opioids to propofol potentiates the risk of postinduction hypotension. Furthermore, opioids increase the risk of postoperative delirium in elderly patients and this risk is further increased with intraoperative hypotension.

Lidocaine is a local anesthetic drug with multiple systemic uses. Lidocaine was proposed to have an anesthetic sparing effect. Lidocaine was previously reported to enhance the hypnotic effect of thiopentone, propofol, and midazolam during procedural sedation. Lidocaine/ketamine combination showed favorable hemodynamic profile following rapid-sequence induction of anesthesia in septic shock patients. Therefore, the use of lidocaine as an adjuvant to propofol might provide a stable cardiovascular profile during induction of anesthesia in elderly compared to fentanyl. To the best of our knowledge, there is no previous data comparing the efficacy of adding lidocaine versus fentanyl to the induction of anesthesia with propofol in elderly

DETAILED DESCRIPTION:
Upon arrival to the operating room, patient's airway will be assessed by trained anesthetist (modified Mallampati test, mouth opening, jaw protrusion, thyromental height, neck extension, dentation). If the patient is considered to be difficult and alternative device other than endotracheal tube is considered, the patients will be excluded. Routine monitors (electrocardiogram, pulse oximetry, and non-invasive blood pressure monitor) will be applied; intravenous line will be secured, and routine pre-medications {ranitidine 50 mg, dexamethasone 4 mg (0.5 mg/ml slow I.V injection)} will be administrated. Baseline preoperative blood pressure will be recorded form the preoperative visit in the supine position as average of 3 readings with difference less than 5 mmHg.

Before induction of anesthesia for all study patients, Electrical cardiometry device (ICON; Cardiotonic, Osypka; Berlin, Germany) will be applied to the patient through 4 electrodes at the following sites: Below the left ear, Above the midpoint of the left clavicle, Left mid-axillary line at level of the xiphoid process and 5 cm inferior to the third electrode. Stroke volume variability (SVV) was measured while patient maintaining standard calm breathing at 8 breath/minute for one-minute. Patients with SVV ≥ 13% will be considered fluid responder and will receive a fluid bolus of 8 mL/kg Ringer acetate over 10 minutes. The fluid bolus will be repeated until the SVV is less than 13%.

Patients will be allocated into two groups: lidocaine group and fentanyl group. In all patients, propofol will be injected slowly in 0.25 mg/kg increments every 20 s till clinical loss of consciousness or reaching a maximum dose of 1-1.5 mg/kg in addition to the study drug. Clinical loss of consciousness (defined as no response to auditory command and disappearance of a patient's eyelash reflex) will be assessed by asking the patients repeatedly every 10 s to open their eyes, when there is no response to auditory commands, the eyelid reflex will be tested. After loss of consciousness, rocuronium (0.6 mg/kg) will be administered, and anesthesia will be maintained by isoflurane (0.9-1% end-tidal). Endotracheal tube will be inserted after 2-minutes of mask ventilation. Ringer lactate solution will be infused at a rate of 2 mL/kg/hour. If the patient did not achieve adequate hypnosis, an additional bolus of propofol (0.5 mg/kg) will be administered.

Any episode of hypotension (defined as mean arterial pressure ≤ 70% of the baseline reading and/or mean arterial pressure <60 mmHg) will be managed by 5 mcg norepinephrine (which can be repeated if hypotension persisted for 2 minutes).

Severe post-induction hypotension defined as mean arterial pressure ≤60% of baseline, will be managed by 5 mcg norepinephrine and the blood pressure will be measure at 1-min interval. Norepinephrine bolus will be repeated if severe hypotension persisted for 1-minute.

If bradycardia occurred (defined as heart rate less than 45 bpm), it will be managed by IV atropine bolus (0.5 mg).

After skin incision, hemodynamic and anesthetic management will be according to the attending anesthetist discretion.

Postoperative Confusion assessment method (CAM) assessment will be performed by trained research member at and 24- and 48-hours after surgery. CAM will be assessed through a four-step algorithm identifying the following: 1) acute onset of mental status changes or a fluctuating course, 2) inattention, 3) disorganized thinking, 4) an altered level of consciousness. Patients will be diagnosed to be delirious if both features {(1) and (2)} will be present plus either feature (3) or (4)}

ELIGIBILITY:
Inclusion Criteria:

* American society of anesthesiologists I-III,
* scheduled for elective non-cardiac surgery under general anesthesia

Exclusion Criteria:

* Patients with severe cardiac morbidities (impaired contractility with ejection fraction < 50%, heart block, arrhythmias, tight valvular lesions, metabolic equivalent less than 4),
* patients on angiotensin converting enzyme inhibitors and angiotensin receptor blockers medications,
* patients with uncontrolled hypertension,
* patients with body mass index <18 or > 35 Kg/m2,
* patient with allergy of any of the study drugs

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
total norepinephrine dose | 1 minute after induction of anesthesia until 15 minutes after induction or surgical incision
  mcg

SECONDARY OUTCOMES:
Incidence of post-induction hypotension | 1 minute after induction of anesthesia until 15 minutes after induction or surgical incision
  mean arterial pressure ≤70% of baseline or < 60 mmHg
Incidence of severe post-induction hypotension | 1 minute after induction of anesthesia until 15 minutes after induction or surgical incision
  mean arterial pressure ≤60% of baseline
Incidence of hypertension | 1 minute after induction of anesthesia until 15 minutes after induction or surgical incision
  mean arterial pressure 120% of baseline
tachycardia | 1 minute after induction of anesthesia until 15 minutes after induction or surgical incision
  heart rate >120% of baseline
loss consciousness time | 1 second after starting drug injection until one second after loss of consciousness
  time to achieve no response to auditory command and disappearance of a patient's eyelash reflex
total propofol dose | 1 second after starting drug injection until one second after loss of consciousness
  mg/kg
intubation time | 1 second after insertion of direct laryngoscopy into the mouth till one second after its removal after tracheal intubation
  second
incidence of postoperative delirium | at 24 and 48 hour postoperatively
  Confusion assessment method will be assessed through a four-step algorithm identifying the following: 1) acute onset of mental status changes or a fluctuating course, 2) inattention, 3) disorganized thinking, 4) an altered level of consciousness. Patients will be diagnosed to be delirious if both features {(1) and (2)} will be present plus either feature (3) or (4)}

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alaini Hospital, Cairo, Egypt